CLINICAL TRIAL: NCT01001091
Title: AL-38583 Ophthalmic Solution for Allergic Conjunctivitis Associated Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Ophthalmic Research Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-034
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Allergic Conjunctivitis
Keywords: Conjunctivitis; conjunctival inflammation; ocular allergies
MeSH Terms: conditions — Conjunctivitis, Allergic; Conjunctivitis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- AL-38583 0.01% (Experimental): AL-38583 ophthalmic solution, 1 drop instilled in each eye 3 times per day for 2 weeks
  Interventions: Drug: AL-38583 ophthalmic solution
- AL-38583 0.05% (Experimental): AL-38583 ophthalmic solution, 1 drop instilled in each eye 3 times per day for 2 weeks
  Interventions: Drug: AL-38583 ophthalmic solution
- AL-38583 0.2% (Experimental): AL-38583 ophthalmic solution, 1 drop instilled in each eye 3 times per day for 2 weeks
  Interventions: Drug: AL-38583 ophthalmic solution
- AL-38583 Vehicle (Placebo Comparator): AL-38583 ophthalmic solution vehicle, 1 drop instilled in each eye 3 times per day for 2 weeks
  Interventions: Drug: AL-38583 ophthalmic solution vehicle
- MAXIDEX (Active Comparator): Dexamethasone ophthalmic suspension, 0.1%, 1 drop instilled in each eye 3 times per day for 2 weeks
  Interventions: Drug: Dexamethasone ophthalmic suspension, 0.1%

INTERVENTIONS:
Drug: AL-38583 ophthalmic solution
  Arms: AL-38583 0.01%; AL-38583 0.05%; AL-38583 0.2%
Drug: AL-38583 ophthalmic solution vehicle — Inactive ingredients used as a placebo comparator
  Arms: AL-38583 Vehicle
Drug: Dexamethasone ophthalmic suspension, 0.1%
  Other Names: MAXIDEX
  Arms: MAXIDEX

SUMMARY:
The purpose of this study is to assess the safety and efficacy of AL-38583 in the treatment of the signs of inflammation associated with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of signs and symptoms of ocular inflammation in both eyes.
* Have a positive CAC response at Visit 1.
* Able to avoid the use of disallowed medications as well as contact lens wear for the specified period prior to Visit 1, and for the duration of the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Have known history or presence of persistent dry eye syndrome.
* Presence of any ophthalmic abnormality that may affect the study outcomes.
* Have a history of moderate to severe allergic asthma reaction to mountain cedar or the perennial allergens used in the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mean area under the curve 0-7 hours post-CAC for conjunctival redness scores | Day 14

SECONDARY OUTCOMES:
Mean daily diary ocular redness scores | 2 week period between Day 0 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Michela Palmer, Study Director — Alcon Research